CLINICAL TRIAL: NCT01529502
Title: Effects of Stored Red Blood Cell Transfusion in Overweight Subjects With Endothelial Dysfunction: Influence of Inhaled Nitric Oxide (iNO)
Brief Title: Pilot Study About the Harmful Effects of Blood Storage on Overweight People and the Role of iNO in This Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Warren M. Zapol, Emeritus Anesthetist-in-Chief and Director of the MGH Anesthesia Center for Critical Care Research, Massachusetts General Hospital; Reginald Jenney Professor of Anesthesia, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Blood Study Overweight
Record Dates: First submitted 2012-02-06; First posted 2012-02-08 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Blood Transfusion; Endothelial Physiopathology; Nitric Oxide; Pulmonary Hypertension
Keywords: Blood Transfusion, Autologous; Blood Preservation/adverse effects; Blood Transfusion/adverse effects; Endothelium, Vascular/physiopathology; Hemoglobins; Nitric Oxide; Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Inosine; Organization and Administration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fresh blood (Experimental)
  Interventions: Procedure: Red blood Cells auto-transfusion
- Old blood (Experimental)
  Interventions: Procedure: Red blood Cells auto-transfusion
- Old blood + inhaled Nitric Oxide (Experimental)
  Interventions: Procedure: Red blood Cells auto-transfusion; Drug: Inhaled Nitric Oxide (iNO) administration

INTERVENTIONS:
Procedure: Red blood Cells auto-transfusion — Withdrawal from 14 overweight volunteers of one unit of red blood cells and auto-transfusion after 3 days storage time. The same 14 subjects will be included in every arm of the study.
  Arms: Fresh blood
Procedure: Red blood Cells auto-transfusion — Withdrawal from the same 14 overweight volunteers of one unit of red blood cells and auto-transfusion after 40 days storage time.
  Arms: Old blood; Old blood + inhaled Nitric Oxide
Drug: Inhaled Nitric Oxide (iNO) administration — Subjects will breath iNO (80ppm) for 10 minutes before, during and for one hour after the autologous old-blood transfusion.
  Arms: Old blood + inhaled Nitric Oxide

SUMMARY:
The purpose of this study is to determine whether storage time affects how human body responds to autologous blood transfusion. An autologous blood transfusion is when a person donates blood and then receives that same blood back in the transfusion. We also want to find out if in this situation inhaled nitric oxide can help to prevent the potential reduction of vasodilation capacity. Vasodilation capacity is the ability of the blood vessel to widen when needed.

DETAILED DESCRIPTION:
The objective of this study is to assess effects of the storage of PRBC on pulmonary vasoconstriction measured as increase in pulmonary artery pressure and endothelial function measured as a change in reactive hyperemia index in overweight people with existing endothelial dysfunction at baseline.

The present study consists of three different parts, which will be scheduled in a randomized order on the same subject (crossover study).

During one phase of the study, 14 healthy human volunteers will donate a unit of Packed Red Blood Cells (PRBC), which will be leukoreduced and stored in Additive Solutions-1 (AS-1), and then transfused back to the subjects after 3 days of storage at 4º C in the MGH Blood Bank (Fresh Blood arm). The second part of the study consists in the collection of another unit of PRBC from the same volunteers which will be transfused back to them after 40 days of storage (Old Blood arm). Finally in the third part, like in the second one, one unit of PRBC will be withdraw and stored for 40 days, but 80 ppm (parts per million by volume) Nitric Oxide in air will be administered together with the transfusion. There will be a 2 weeks interval after each PRBC transfusion.

We hypothesize that old red blood cells stored under conventional conditions may trigger a complex, pro-inflammatory, pro-thrombotic and vasoconstriction response. We will compare the response to PRBC stored for 3 days with the response to PRBC stored for 40 days in the same healthy volunteers. We also want to test the hypothesis that inhaled nitric oxide may reverse these adverse effects.

We will monitor/measure the following parameters:

1. Pulmonary vasoconstriction by trans-thoracic echocardiography
2. Endothelium-mediated changes in vascular (arterial) tone, measured as reactive hyperemia index.

ELIGIBILITY:
Inclusion Criteria:

1. Have a photo ID
2. Age>18 years old (required to provide informed consent)
3. Age <60 years old
4. Mild impairment of endothelial function, assessed by post ischemic vasodilation (L_RHI,<0.7) (38)
5. Body mass index (BMI) >27 kg/m^2 and <40 kg/m^2
6. Fasting during the days of transfusion.
7. Avoiding intake of high nitrate food (i.e. green leafy vegetables: lettuce, spinach) on the day prior to the study
8. Feel well on the day of blood donation
9. KG within normal limits
10. Normotensive (systolic blood pressure <140 mmHg and diastolic <90 mmHg)
11. Normal physical exam and blood test results as indicated by:

    1. WBC 4.5-11.0 n x103/μL
    2. HGB 12.0-17.5 gm/dl
    3. PLT 150-400 n x103/μL
    4. Plasma Sodium 135-145 mmol/L
    5. Plasma Potassium 3.4-4.8 mmol/L
    6. Plasma Chloride 98-108 mmol/L
    7. Plasma Carbon Dioxide 23.0-31.9 mmol/L
    8. Plasma Urea Nitrogen 8-25 mg/dl
    9. Plasma Creatinine 0.60-1.50 mg/dl
    10. Plasma Glucose 70-110 mg/dl
    11. Transaminase-SGPT 10-55 U/L
    12. Transaminase-SGOT 10-40 U/L
    13. Total Bilirubin < 2 mg/dl
    14. Fasting plasma glucose < 110 mg/dl
    15. Methemoglobin < 3%

Exclusion Criteria:

1. Psychiatric disturbances such as anxiety, depression, schizophrenia requiring pharmacological treatment or hospitalization in the last year
2. Systemic disease with or without any functional limitation
3. Pregnancy determined by urine pregnancy test, detecting presence of human chorionic gonadotropin (hCG), or less than six weeks postpartum
4. Active smoking. Volunteers may be enrolled if they quit smoking for more than 1 year.
5. Excess alcohol use: more than ½ L/day of wine consumption or equivalent
6. Any current use of a medication other than: over-the-counter oral medications, herbal remedies, nutritional supplements, and oral contraceptives.
7. Antibiotic use within 48 hours of blood donation
8. Use of NSAIDS, corticosteroids, aspirin during the past 7 days
9. Dental work within 24 hours prior to the donation
10. Received or donated blood in the last 4 months
11. Have had any forms of cancer with the exceptions of basal cell skin cancer or treatment for in situ uterine cervical cancer
12. Currently enrolled in another research study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren Zapol, MD, Principal Investigator — Masachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hendrickson JE, Hillyer CD. Noninfectious serious hazards of transfusion. Anesth Analg. 2009 Mar;108(3):759-69. doi: 10.1213/ane.0b013e3181930a6e. PMID 19224780
- [Background] Koch CG, Li L, Sessler DI, Figueroa P, Hoeltge GA, Mihaljevic T, Blackstone EH. Duration of red-cell storage and complications after cardiac surgery. N Engl J Med. 2008 Mar 20;358(12):1229-39. doi: 10.1056/NEJMoa070403. PMID 18354101
- [Background] Bennett-Guerrero E, Veldman TH, Doctor A, Telen MJ, Ortel TL, Reid TS, Mulherin MA, Zhu H, Buck RD, Califf RM, McMahon TJ. Evolution of adverse changes in stored RBCs. Proc Natl Acad Sci U S A. 2007 Oct 23;104(43):17063-8. doi: 10.1073/pnas.0708160104. Epub 2007 Oct 11. PMID 17940021
- [Background] Cardillo C, Kilcoyne CM, Cannon RO 3rd, Panza JA. Interactions between nitric oxide and endothelin in the regulation of vascular tone of human resistance vessels in vivo. Hypertension. 2000 Jun;35(6):1237-41. doi: 10.1161/01.hyp.35.6.1237. PMID 10856270
- [Background] Panza JA, Casino PR, Kilcoyne CM, Quyyumi AA. Role of endothelium-derived nitric oxide in the abnormal endothelium-dependent vascular relaxation of patients with essential hypertension. Circulation. 1993 May;87(5):1468-74. doi: 10.1161/01.cir.87.5.1468. PMID 8491001
- [Background] Hod EA, Brittenham GM, Billote GB, Francis RO, Ginzburg YZ, Hendrickson JE, Jhang J, Schwartz J, Sharma S, Sheth S, Sireci AN, Stephens HL, Stotler BA, Wojczyk BS, Zimring JC, Spitalnik SL. Transfusion of human volunteers with older, stored red blood cells produces extravascular hemolysis and circulating non-transferrin-bound iron. Blood. 2011 Dec 15;118(25):6675-82. doi: 10.1182/blood-2011-08-371849. Epub 2011 Oct 20. PMID 22021369
- [Derived] Berra L, Pinciroli R, Stowell CP, Wang L, Yu B, Fernandez BO, Feelisch M, Mietto C, Hod EA, Chipman D, Scherrer-Crosbie M, Bloch KD, Zapol WM. Autologous transfusion of stored red blood cells increases pulmonary artery pressure. Am J Respir Crit Care Med. 2014 Oct 1;190(7):800-7. doi: 10.1164/rccm.201405-0850OC. PMID 25162920

RESULTS

PARTICIPANT FLOW:
Groups:
- Fresh Blood - Old Blood - Old Blood+iNO; Old Blood - Fresh Blood - Old Blood+iNO; Old Blood+iNO - Old Blood - Fresh Blood; Fresh Blood - Old Blood+iNO - Old Blood; Old Blood - Old Blood+iNO - Fresh Blood; Old Blood+iNO - Fresh Blood - Old Blood: FRESH BLOOD:
  Red blood Cells auto-transfusion: Withdrawal from same overweight volunteers of one unit of red blood cells and auto-transfusion after 3 days storage time.
  OLD BLOOD:
  Red blood Cells auto-transfusion: Withdrawal from same overweight volunteers of one unit of red blood cells and auto-transfusion after 40 days storage time.
  OLD BLOOD+iNO Red blood Cells auto-transfusion: Withdrawal from same overweight volunteers of one unit of red blood cells and auto-transfusion after 40 days storage time while breathing Nitric Oxide (NO).
Period: Overall Study
Arm/Group | Fresh Blood - Old Blood - Old Blood+iNO | Old Blood - Fresh Blood - Old Blood+iNO | Old Blood+iNO - Old Blood - Fresh Blood | Fresh Blood - Old Blood+iNO - Old Blood | Old Blood - Old Blood+iNO - Fresh Blood | Old Blood+iNO - Fresh Blood - Old Blood
Started | 2 | 3 | 2 | 3 | 2 | 2
Completed | 2 | 3 | 2 | 1 | 2 | 2
Not Completed | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fresh Blood-Old Blood-Old Blood + Inhaled Nitric Oxide; Fresh Blood-Old Blood + Inhaled Nitric Oxide-Old Blood-; Old Blood- Fresh Blood- Old Blood + Inhaled Nitric Oxide; Old Blood- Old Blood + Inhaled Nitric Oxide- Fresh Blood; Old Blood + Inhaled Nitric Oxide- Fresh Blood- Old Blood; Old Blood + Inhaled Nitric Oxide- Old Blood- Fresh Blood: FRESH BLOOD:
  Red blood Cells auto-transfusion: Withdrawal from the same overweight volunteers of one unit of red blood cells and auto-transfusion after 3 days storage time.
  OLD BLOOD:
  Red blood Cells auto-transfusion: Withdrawal from the same overweight volunteers of one unit of red blood cells and auto-transfusion after 40 days storage time.
  OLD BLOOD + inhaled NITRIC OXIDE Red blood Cells auto-transfusion: Withdrawal from the same overweight volunteers of one unit of red blood cells and auto-transfusion after 40 days storage time.
  Inhaled Nitric Oxide (iNO) administration: Subjects will breath iNO (80ppm) for 10 minutes before, during and for one hour after the autologous old-blood transfusion.
- Total: Total of all reporting groups
Arm/Group | Fresh Blood-Old Blood-Old Blood + Inhaled Nitric Oxide | Fresh Blood-Old Blood + Inhaled Nitric Oxide-Old Blood- | Old Blood- Fresh Blood- Old Blood + Inhaled Nitric Oxide | Old Blood- Old Blood + Inhaled Nitric Oxide- Fresh Blood | Old Blood + Inhaled Nitric Oxide- Fresh Blood- Old Blood | Old Blood + Inhaled Nitric Oxide- Old Blood- Fresh Blood | Total
Number analyzed (Participants) | 2 | 3 | 3 | 2 | 2 | 2 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 3 | 2 | 2 | 2 | 14
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 46 [30 to 64] | 37 [22 to 46] | 46 [34 to 60] | 26.5 [26 to 27] | 51 [49 to 53] | 41 [29 to 53] | 41 [22 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 1 | 1 | 1 | 5
  Male | 2 | 2 | 2 | 1 | 1 | 1 | 9
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 3 | 2 | 2 | 2 | 14
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 37 [33 to 40] | 33 [28 to 37] | 30 [28 to 31] | 33.5 [32 to 35] | 35.5 [31 to 40] | 33 [31 to 35] | 33 [28 to 40]

OUTCOME MEASURES:

1. Primary Outcome: Systolic Pulmonary Artery Pressure
Description: Pulmonary vasoconstriction was measured by estimation of Systolic Pulmonary Artery Pressure in millimeter of mercury (mmHg) by trans-thoracic echocardiography
Time Frame: Post-transfusion
Population: In the "fresh blood" only 9 volunteers estimation of Systolic Pulmonary Artery Pressure was successfully studied by trans-thoracic echocardiography. In the "old blood" only 11 volunteers and In the "old blood + Inhaled Nitric Oxide" only 12 volunteers estimation of Systolic Pulmonary Artery Pressure was successfully evaluated.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Fresh Blood | Old Blood | Old Blood + Inhaled Nitric Oxide
Number analyzed (Participants) | 9 | 11 | 12
mmHg | 39 (3) | 46 (3) | 31 (2)

2. Secondary Outcome: Endothelial Function: Reactive Hyperemia Index
Description: Reactive Hyperemia Index (RHI) measures Endothelial function and is assessed by digital pulse amplitude tonometry and it is a sensitive indicator of endothelial function. RHI is a calculated as a ratio between tested versus contralateral finger dilatation, thus there is no unit measure.
Time Frame: Post-transfusion
Measure: Mean (Standard Error); unit: LnRHI
Arm/Group | Fresh Blood | Old Blood | Old Blood + Inhaled Nitric Oxide
Number analyzed (Participants) | 9 | 11 | 12
LnRHI | 0.87 (0.06) | 0.9 (0.06) | 0.78 (0.06)

3. Other Pre Specified Outcome: Hemolysis
Description: To assess concentration of plasma Hemoglobin at baseline, 10 minutes after blood transfusion, 1 hour after blood transfusion, 2 hours after blood transfusion and 4 hours after blood transfusion.
Time Frame: before and after blood transfusion
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Nitric Oxide Metabolites
Description: To assess concentration of plasma Nitric oxide metabolites at baseline, 10 minutes after blood transfusion, 1 hour after blood transfusion, 2 hours after blood transfusion and 4 hours after blood transfusion.
Time Frame: Before and after blood transfusion
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Concentration of Cytokines
Description: To assess concentration of plasma cytokines at baseline, 10 minutes after blood transfusion, 1 hour after blood transfusion, 2 hours after blood transfusion and 4 hours after blood transfusion.
Time Frame: Before and after blood transfusion
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Activation of Platelets
Description: To assess concentration of plasma activation of platelets at baseline, 10 minutes after blood transfusion, 1 hour after blood transfusion, 2 hours after blood transfusion and 4 hours after blood transfusion.
Time Frame: Before and after blood transfusion
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Activation of Inflammatory Lipid Mediators
Description: To assess concentration of plasma activation of inflammatory lipid mediators at baseline, 10 minutes after blood transfusion, 1 hour after blood transfusion, 2 hours after blood transfusion and 4 hours after blood transfusion.
Time Frame: Before and after blood transfusion
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Changes in Gene Expression
Description: To assess concentration of changes in gene expression at baseline, 10 minutes after blood transfusion, 1 hour after blood transfusion, 2 hours after blood transfusion and 4 hours after blood transfusion.
Time Frame: Before and after blood transfusion
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Endothelial Function
Description: To assess Endothelial function by RHI at baseline, 10 minutes after blood transfusion, 1 hour after blood transfusion, 2 hours after blood transfusion and 4 hours after blood transfusion.
Time Frame: Before and after blood transfusion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Time over which adverse event data were collected was during blood transfusion up to 1 day after transfusion
Description: 14 volunteers were enrolled in the study and received the "Fresh Blood". Two of the 14 volunteers left the study before finishing all three arms. One of the two of the volunteers that left the study, completed the "Fresh Blood" and "Old Blood", thus 13 volunteers completed the "Old Blood" arm. The last volunteer left before receiving "Old Blood + Inhaled Nitric Oxide", thus the number of participants in and the the "Old Blood + Inhaled Nitric Oxide" arm is twelve.
Arm/Group | Fresh Blood | Old Blood | Old Blood + Inhaled Nitric Oxide
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes